CLINICAL TRIAL: NCT06623318
Title: IV Ensure in Patients Receiving OPAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IV Ensure (Industry)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IVEnsure
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Determine If Adherence Rates with IV Antibiotics in OPAT Have a Correlation to Hospital Readmission Rates
Keywords: OPAT; IV antibiotic; Adherence; home infusion; readmission

STUDY DESIGN:
Intervention Model Description: The investigation will be designed as a retrospective cohort study, in which assignment to the IV Ensure device is determined based on patient discharge status (home IV for antimicrobial therapy) and current device allocation. Patients will be assigned to IV Ensure subsequent to their initial health encounter for their admitting diagnosis. The non-treatment group will be assigned to home infusion therapy using the current standard of care of OU Medicine. This group is required in order to assess whether the usage of the IV Ensure device is associated with a reduction in subsequent readmission risk due to infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Determine adherence rate for IV medications administered in the home. (Experimental): Patients will be assigned IV Ensure's remote therapeutic monitoring device to determine their adherence rate with administration of IV medications administered in the home in comparison to their provider's orders.
  Interventions: Device: Remote therapeutic monitoring device
- Assess re-admission against adherence rates. (Experimental): Assess correlation of patients hospital re-admission rates for infection related disease progression associated with adherence rates of IV medications administered in the home.
  Interventions: Device: Remote therapeutic monitoring device

INTERVENTIONS:
Device: Remote therapeutic monitoring device — IV Ensure proprietary remote therapeutic monitoring device is used to record and transmit data associated with date, time, and duration of IV medications administered in the home setting post-acute.
  Other Names: IV Advocate

SUMMARY:
The purpose of remote therapeutic monitoring is to provide oversight and evaluation of patients receiving IV medications in the home setting post-acute. The goal is to improve patient outcomes and decrease re-admission rates for related diagnoses due to poor adherence. Remote therapeutic monitoring provides data used in the determination of dates, times, and duration of doses administered in the home setting to support real-time intervention by dedicated care managers to support improved adherence with prescribed dosing regiments. The objectives of the study are to:

1. Determine adherence rates for IV medications administered in the home.
2. Assess re-admission against adherence rates.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients enrolled in OPAT (IV antibiotic therapy) discharged to the home setting will be included in the study.

Exclusion Criteria:

* Patients enrolled in OPAT (IV antibiotic therapy) discharged to nursing homes, SNF (Skilled Nursing Facility), and pediatric patients will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Readmission due to subsequent related infection following the initial encounter. | From enrollment to 30 days after completion of prescribed IV medication.
  This will be defined as a dichotomous outcome variable with Yes occurring when (a) a patients ID reoccurs in the OU Medicine EMR/EHR data pull within 30 days of their discharge with IV Ensure remote therapeutic monitoring device and (b) the patients readmissions reason matched the pre-specified list of ICD codes corresponding to secondary or downstream infections. If both of the above do not occur, the readmission variable will be set to No.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sassine, MD, FACP, Principal Investigator — The University of Oklahoma Health Sciences Center
Locations (1):
- The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
The participant information will not be used or distributed for future research studies.